CLINICAL TRIAL: NCT04134676
Title: Therapeutic Potential of Stem Cell Conditioned Medium on Chronic Ulcer Wounds : Pilot Study in Human
Brief Title: Therapeutic Potential of Stem Cell Conditioned Medium on Chronic Ulcer Wounds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sukma Skin Treatment (Other)
Collaborators: Stem Cell and Cancer Institute, Kalbe Farma Tbk (Unknown); PT Pharma Metric Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PML-KLB-02-2019
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Chronic Ulcer
Keywords: Stem Cell; Conditioned Medium
MeSH Terms: interventions — Culture Media, Conditioned

STUDY DESIGN:
Intervention Model Description: Experimental clinical trial with open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conditioned Medium Group (Experimental): In this group, the subjects will use Conditioned Medium topical therapy for 2 weeks The Conditioned Medium gel will be applied to the wound and closed by transparent dressing.
  The evaluation and dressing replacement will be done every week for 2 weeks.
  Interventions: Drug: Conditioned Media

INTERVENTIONS:
Drug: Conditioned Media — Conditioned Media represents the complete regenerative milieu of cell-sourced secretome and vesicular elements. The soluble components of the secretome may be separated from the microvesicle fraction by centrifugation, filtration, polymer precipitation-based methodologies, ion exchange chromatography and size-exclusion chromatography. Both of these components may be capable of independently triggering regeneration and repair as well as of mediating the de novo organogenesis of tissue-engineered organs ex vivo.

SUMMARY:
Chronic wounds (CW) still represents a heavy burden to many patients and health care institution. Despite the most recent advances in wound management, up to 50% of chronic wounds still fail to heal. Conventional treatment of chronic wounds does not seem to work in several cases, consumes enormous amount of money and time, so it is necessary to develop different strategies. Previous studies have reported stem cells ability in tissue regenerations due mainly to its secreted paracrine factors, rather than its differentiation ability to become new cells. The factors is called secretomes, microvesicles, or exosomes, that can be found in the medium where the cells are growing, therefore it called conditioned medium (CM). Mesenchymal stem cells (MSCs) such as Wharton's Jelly Mesenchymal Stem Cells (WJ-MSC) appear to emerge as a promising wound healing therapy. To the best of investigator's knowledge, after conducted a pilot study using animal model to gain the preliminary data for the ulcer healing potential, this is the investigator's first clinical study to see the therapeutic potentials of Conditioned Medium Stem Cell as an additional growth factors in chronic skin ulcer healing and to compare the success of chronic ulcer healing in patients undergoing CM treatment and standard approach. The investigators will examine the therapeutic effect of human WJ-MSC-CM in wound healing on patients with chronic skin ulcer.

DETAILED DESCRIPTION:
Treatment for chronic wound healing has become a great challenge in medical world. The incidence of chronic non healing wounds continues to increase and the classical method for wound healing therapy no longer reliable for chronic wounds healing. Therefore a new alternative strategy to control chronic wound healing is needed. Stem cell therapy has become a leading alternative strategy for wound healing therapy in this new modern world. The development of using conditioned medium such as Wharton's Jelly Mesenchymal Stem Cells have arising because of its paracrine factors that can provide a better healing process. During daily practice at the clinic, the authors sometimes find patients with chronic skin ulcers that cannot be treated using standard therapy. This encourages the authors to innovate new therapy to help the wound healing process by using human WJ-MSC conditioned medium.

This study has several purposes, such as; to observe the success rate, the differences in the period of time needed, and the differences in wound closure of chronic ulcer healing in patients undergoing wound care with conditioned medium and standard therapy. As for the benefits of research, these are the benefits; reducing the cost spent on treatment in chronic skin ulcer, faster chronic wound healing while minimizing the complications, improving the quality of therapy for patients with chronic skin ulcers, reducing the treatment period for chronic skin ulcer and can be used as the basis for future researchers to conduct further research on Conditioned Medium Stem Cell and chronic wound management.

Stem cell therapy constitutes a new alternative methods of wound healing. Many researchers are relying on this alternative new therapy that holds great potentials for its growth factors. Mesenchymal stem cell (MSCs) have been isolated from many types of adult tissues and fetal tissues, such as umbilical cord, skin, and placenta. When engrafted at sites of tissue injury, MSCs differentiate into connective tissue elements, support vasculogenesis, and secretes cytokines and growth factors that facilitate healing. As in wounds, MSCs differentiate into fibroblasts and pericytes and, perhaps, endothelial-like or vessel attached cells. WJ-MSCs secrete proangiogenic and wound healing promoting factors, such as transforming growth factor beta (TGF-β), vascular endothelial growth factor (VEGF), platelet-derived growth factor, insulin-like growth factor-I, interleukin (IL)-6 and IL-8.

The use of MSC-sourced secretome in regenerative medicine provides key advantages over stem-cell based applications such as; (a) resolving several safety considerations potentially associated with the transplantation of living and proliferative cell populations, (b) can be evaluated for safety, dosage and potency, (c) storage can be done without application of potentially toxic cryopreservative agents for a long period without loss of product potency, (d) using MSC-sourced secretome, such as conditioned medium (CM), is more economical and more practical for clinical application since it avoids invasive cell collection procedures, (e) the time and cost of expansion and maintenance of cultured stem cells could be greatly reduced, (f) finally, the biological product obtained for therapeutic applications could be modified to desired cell-specific effects.

This research is an experimental clinical trial with open label. This research will be conducted in Sitanala Village (RW 001), Mayapada Hospital, Indra Clinic and Sukma Clinic, Banten. Conditioned Medium Stem Cell obtained from SCI (PT. Kalbe Farma, Tbk.). The study started from June 2019 to June 2020. The sample used from this study are all outpatient and hospitalized patients with chronic skin ulcers at Mayapada Hospital, Indra Clinic, Sukma Clinic and Sitanala Village (RW 001) from June 2019 until May 2020. In this pilot study, 38 subjects will be included based on estimated sample size. The method of selecting samples is by using consecutive sampling. Data was collected by measuring the first ulcer and taking photos of each subject. The patient then use CM topical therapy and the evaluation is carried out after 2 weeks. Results are expressed as means ± SD. The normal distribution of the data was assessed using the Shapiro-Wilk test. For multiple comparisons One-Way Analysis of Variance (ANOVA) was used. The significance between two independent groups was determined by independent Student's t-test and the Mann-Whitney test. An unpaired t-test was performed if the data were normally distributed. Otherwise, a Mann-Whitney test was used. Statistical analysis was 2-tailed and values were considered statistically significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic skin ulcer that had received therapy for more than 1 month but there were no improvements

Exclusion Criteria:

* Respondent who refused to be the subject of this research
* ulcer size >10 x 15 cm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Knowing the the success rate of chronic ulcer healing in patients undergoing wound care with conditioned medium | The ulcer is measured after 2 weeks
  Assessing ulcer progression macroscopic evaluation of:
  * The presence of granulation tissue
  * The size of the ulcer reduced
  * Edema decreases
  * Erythema decreases
  Results are expressed as means ± SD. The normal distribution of the data was assessed using the Shapiro-Wilk test. For multiple comparisons One-Way Analysis of Variance (ANOVA) was used. The significance between two independent groups was determined by independent Student's t-test and the Mann-Whitney test. An unpaired t-test was performed if the data were normally distributed. Otherwise, a Mann-Whitney test was used. Statistical analysis was 2-tailed and values were considered statistically significant at p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Sukmawati T Tan, Dr. dr., Principal Investigator — Tarumanagara University; Siufui Hendrawan, Dr. dr, Study Director — Tarumanagara University
Locations (3):
- Indonesia (3):
  - Mayapada Hospital, Tangerang, Banten
  - Indra Clinic, Tangerang, Banten
  - Sukma Cliniq, Tangerang, Banten

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Chen J, Kirsner R. Pathophysiology of acute wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):9-18. doi: 10.1016/j.clindermatol.2006.09.007. PMID 17276196
- [Background] de la Garza-Rodea AS, Knaan-Shanzer S, van Bekkum DW. Pressure ulcers: description of a new model and use of mesenchymal stem cells for repair. Dermatology. 2011;223(3):266-84. doi: 10.1159/000334628. Epub 2011 Nov 23. PMID 22116308
- [Background] Posnett J, Franks PJ. The burden of chronic wounds in the UK. Nurs Times. 2008 Jan 22-28;104(3):44-5. PMID 18293879
- [Background] Turner NJ, Badylak SF. The Use of Biologic Scaffolds in the Treatment of Chronic Nonhealing Wounds. Adv Wound Care (New Rochelle). 2015 Aug 1;4(8):490-500. doi: 10.1089/wound.2014.0604. PMID 26244105
- [Background] Bluestein D, Javaheri A. Pressure ulcers: prevention, evaluation, and management. Am Fam Physician. 2008 Nov 15;78(10):1186-94. PMID 19035067
- [Background] Xu Y, Guo S, Wei C, Li H, Chen L, Yin C, Zhang C. The Comparison of Adipose Stem Cell and Placental Stem Cell in Secretion Characteristics and in Facial Antiaging. Stem Cells Int. 2016;2016:7315830. doi: 10.1155/2016/7315830. Epub 2016 Feb 8. PMID 27057176
- [Background] Arno AI, Amini-Nik S, Blit PH, Al-Shehab M, Belo C, Herer E, Tien CH, Jeschke MG. Human Wharton's jelly mesenchymal stem cells promote skin wound healing through paracrine signaling. Stem Cell Res Ther. 2014 Feb 24;5(1):28. doi: 10.1186/scrt417. PMID 24564987
- [Background] Khosrotehrani K. Mesenchymal stem cell therapy in skin: why and what for? Exp Dermatol. 2013 May;22(5):307-10. doi: 10.1111/exd.12141. PMID 23614735
- [Background] Klopp AH, Gupta A, Spaeth E, Andreeff M, Marini F 3rd. Concise review: Dissecting a discrepancy in the literature: do mesenchymal stem cells support or suppress tumor growth? Stem Cells. 2011 Jan;29(1):11-9. doi: 10.1002/stem.559. PMID 21280155
- [Background] Kim SM, Lim JY, Park SI, Jeong CH, Oh JH, Jeong M, Oh W, Park SH, Sung YC, Jeun SS. Gene therapy using TRAIL-secreting human umbilical cord blood-derived mesenchymal stem cells against intracranial glioma. Cancer Res. 2008 Dec 1;68(23):9614-23. doi: 10.1158/0008-5472.CAN-08-0451. PMID 19047138
- [Background] Beckermann BM, Kallifatidis G, Groth A, Frommhold D, Apel A, Mattern J, Salnikov AV, Moldenhauer G, Wagner W, Diehlmann A, Saffrich R, Schubert M, Ho AD, Giese N, Buchler MW, Friess H, Buchler P, Herr I. VEGF expression by mesenchymal stem cells contributes to angiogenesis in pancreatic carcinoma. Br J Cancer. 2008 Aug 19;99(4):622-31. doi: 10.1038/sj.bjc.6604508. Epub 2008 Jul 29. PMID 18665180
- [Background] Ho J, Walsh C, Yue D, Dardik A, Cheema U. Current Advancements and Strategies in Tissue Engineering for Wound Healing: A Comprehensive Review. Adv Wound Care (New Rochelle). 2017 Jun 1;6(6):191-209. doi: 10.1089/wound.2016.0723. PMID 28616360
- [Background] Sinno H, Prakash S. Complements and the wound healing cascade: an updated review. Plast Surg Int. 2013;2013:146764. doi: 10.1155/2013/146764. Epub 2013 Jul 24. PMID 23984063
- [Background] McDaniel JC, Browning KK. Smoking, chronic wound healing, and implications for evidence-based practice. J Wound Ostomy Continence Nurs. 2014 Sep-Oct;41(5):415-23; quiz E1-2. doi: 10.1097/WON.0000000000000057. PMID 25188797
- [Background] Coleman S, Gorecki C, Nelson EA, Closs SJ, Defloor T, Halfens R, Farrin A, Brown J, Schoonhoven L, Nixon J. Patient risk factors for pressure ulcer development: systematic review. Int J Nurs Stud. 2013 Jul;50(7):974-1003. doi: 10.1016/j.ijnurstu.2012.11.019. Epub 2013 Feb 1. PMID 23375662
- [Background] Sarasua JG, Lopez SP, Viejo MA, Basterrechea MP, Rodriguez AF, Gutierrez AF, Gala JG, Menendez YM, Augusto DE, Arias AP, Hernandez JO. Treatment of pressure ulcers with autologous bone marrow nuclear cells in patients with spinal cord injury. J Spinal Cord Med. 2011;34(3):301-7. doi: 10.1179/2045772311Y.0000000010. PMID 21756569
- [Background] Singh R, Singh R, Rohilla RK, Siwach R, Verma V, Kaur K. Surgery for pressure ulcers improves general health and quality of life in patients with spinal cord injury. J Spinal Cord Med. 2010;33(4):396-400. doi: 10.1080/10790268.2010.11689718. PMID 21061899
- [Background] Cerqueira MT, Pirraco RP, Marques AP. Stem Cells in Skin Wound Healing: Are We There Yet? Adv Wound Care (New Rochelle). 2016 Apr 1;5(4):164-175. doi: 10.1089/wound.2014.0607. PMID 27076994
- [Background] Vizoso FJ, Eiro N, Cid S, Schneider J, Perez-Fernandez R. Mesenchymal Stem Cell Secretome: Toward Cell-Free Therapeutic Strategies in Regenerative Medicine. Int J Mol Sci. 2017 Aug 25;18(9):1852. doi: 10.3390/ijms18091852. PMID 28841158
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Spaeth EL, Dembinski JL, Sasser AK, Watson K, Klopp A, Hall B, Andreeff M, Marini F. Mesenchymal stem cell transition to tumor-associated fibroblasts contributes to fibrovascular network expansion and tumor progression. PLoS One. 2009;4(4):e4992. doi: 10.1371/journal.pone.0004992. Epub 2009 Apr 7. PMID 19352430
- [Background] Short B, Brouard N, Occhiodoro-Scott T, Ramakrishnan A, Simmons PJ. Mesenchymal stem cells. Arch Med Res. 2003 Nov-Dec;34(6):565-71. doi: 10.1016/j.arcmed.2003.09.007. PMID 14734097
- [Background] Choi M, Lee HS, Naidansaren P, Kim HK, O E, Cha JH, Ahn HY, Yang PI, Shin JC, Joe YA. Proangiogenic features of Wharton's jelly-derived mesenchymal stromal/stem cells and their ability to form functional vessels. Int J Biochem Cell Biol. 2013 Mar;45(3):560-70. doi: 10.1016/j.biocel.2012.12.001. Epub 2012 Dec 12. PMID 23246593
- See also: Immune characterization of mesenchymal stem cells in human umbilical cord Wharton's jelly and derived cartilage cells — http://dx.doi.org/10.1016/j.cellimm.2012.06.010